CLINICAL TRIAL: NCT02516956
Title: Impact of Different Breakfast Meals on Food Choices, Eating Behaviors and Brain Activation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Professor Furio Brighenti, Professor, University of Parma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BRNN-014
Record Dates: First submitted 2015-07-31; First posted 2015-08-06 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Regulation, Appetite; Eating Behavior; Cognition
Keywords: Breakfast; Food choices; Lunch; Eating habits; Appetite; Neural activation; Attention; Glucose; Insulin; fMRI
MeSH Terms: conditions — Feeding Behavior; Insulin Resistance | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Breakfast meal 1 (Experimental): Breakfast meal 1 is isocaloric (330 kcal) and similar for protein and fiber contents in relation to the other two experimental breakfasts. It has the same sugar and lipid profiles as Breakfast meal 2 and health-related cognitive perception as Breakfast meal 3.
  Breakfast consumption; Blood tests; Food choices and energy intakes assessments; Attention tests; fRMI tests.
  Interventions: Other: Breakfast consumption; Other: Blood tests; Other: Food choices and energy intakes assessments; Other: Attention tests; Other: fRMI tests
- Breakfast meal 2 (Experimental): Breakfast meal 2 is isocaloric (330 kcal) and balanced for protein and fiber contents with regard to the other two experimental breakfasts. It has the same sugar and lipid profiles as Breakfast meal 1 but a higher health-related cognitive perception than the other two experimental breakfasts.
  Breakfast consumption; Blood tests; Food choices and energy intakes assessments; Attention tests; fRMI tests.
  Interventions: Other: Breakfast consumption; Other: Blood tests; Other: Food choices and energy intakes assessments; Other: Attention tests; Other: fRMI tests
- Breakfast meal 3 (Experimental): Breakfast meal 3 is isocaloric (330 kcal) and similar for protein and fiber contents in relation to the other two experimental breakfasts. It has the same health-related cognitive perception as Breakfast meal 1 but lower lipid and higher sugar amounts than the other two experimental breakfasts.
  Breakfast consumption; Blood tests; Food choices and energy intakes assessments; Attention tests; fRMI tests.
  Interventions: Other: Breakfast consumption; Other: Blood tests; Other: Food choices and energy intakes assessments; Other: Attention tests; Other: fRMI tests
- Breakfast meal 4 (Placebo Comparator): Breakfast meal 4 is a non-caloric meal representing fasting condition (control arm).
  Breakfast consumption; Blood tests; Food choices and energy intakes assessments; Attention tests; fRMI tests.
  Interventions: Other: Breakfast consumption; Other: Blood tests; Other: Food choices and energy intakes assessments; Other: Attention tests; Other: fRMI tests

INTERVENTIONS:
Other: Breakfast consumption — Participants will consume the assigned breakfast each morning for 7 days. Participants will express a hedonic rating of the breakfast through 7-point Likert Scales before (overview) and after breakfast consumption.
Other: Blood tests — On the third day, participants will be involved in blood tests. Blood will be taken at baseline (fasting), and up to 4 hours after consuming the breakfast. Participants will complete serial visual analog rating scales of hunger and fullness before (fasting) and every 30 minutes up to 4 hours after breakfast consumption.
Other: Food choices and energy intakes assessments — Following the last blood sample, participants will be given the opportunity to consume food ad libitum from a buffet lunch. Double weighing of food will be set up to evaluate food choices and energy intake of lunch. During the test week, participants will record all foods and beverage on a 7-day food dairy.
Other: Attention tests — On the fourth day, 4 hours after the breakfast consumption and avoid other foods, participants will be involved in attentional test (Mackworth Clock Test for sustained attention and Stroop Test for selective attention).
Other: fRMI tests — On the fifth day, 4 hours after the breakfast consumption and avoid other foods, participants will focus on a set of photographs (stimuli will be randomly choose from three categories of pictures including food, nonfood, and blurred baseline images) during an fMRI brain scan procedure to scan brain activation responses

SUMMARY:
This project aims to demonstrate that the best breakfast meal is the one able to improve the best postprandial hunger, satiety and adiposity regulators profile as well as the best reward-related gratification, due to hedonistic parameters. To do this, 4 different breakfasts will be tested and blood tests, food choices, and attentional components will be analysed.

DETAILED DESCRIPTION:
Although breakfast seems to be positively associated with healthy eating patterns and food choices later in the day, eating behaviours are a complex interaction of several factors. Nutritional requirements are not only affected by the body homeostasis, but also by environmental signals, as cultural and social habits, lifestyle, etc. These parameters evoke reward-related and motivational signals influencing our daily eating behaviour choices. Most of the theories on food regulation propose two parallel systems interacting with food consumption homeostatic and reward-related systems. For all these reasons, there is an increasing interest on motivational and decisional aspects of food choices, eating behaviours and how they are influenced by food characteristics. This project aims to explore the association between compositional and perceived characteristics of a breakfast meal with nutritional/biochemical/physiological variables. The approach will be the evaluation of appetite, food intake as well as metabolic and compensatory responses to foods consumed during the day. Volunteers (n=15) will be fed with 4 different breakfast meals (one control and three iso-caloric with different glycemic indexes) and several different parameters will be evaluated, as biological parameters linked to satiety, food choices during a free lunch buffet, psycho-physiological and biological mechanisms underlying the compensatory effect and attentional components in the postprandial period. The participants will complete, in randomized order, the four breakfast meals, on four different weeks, separated by at least one week.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* age 19 - 29 y
* BMI 20-24 kg ⁄m2
* healthy
* no metabolic, psychological, or neurological diseases/conditions
* not currently/previously (in the past 6 months) on a weight loss/other special diet
* omnivorous
* chocolate eaters
* right-handed (necessary for the fMRI analyses)

Exclusion Criteria:

* BMI < 20 or BMI > 24 kg ⁄m2
* chronic health conditions
* use of medications
* significant change in body weight in the last 3 months
* currently on a diet/food restriction
* food allergy
* celiac disease
* lactose intolerance
* left-handed
* claustrophobic
* do not meet the fMRI criteria established by the MU-BIC (regarding metal implants, etc.)
* pregnant

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in biomarkers of appetite regulation in response to each breakfast: | 4 hours (0 -12h fasting-, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 minutes)
  * Glucose
  * Insulin
  * Ghrelin
  * Leptin
  * Peptide YY
  * Glucagon-like peptide-1
  * Non Esterified Fatty Acids

SECONDARY OUTCOMES:
Hedonic rating of breakfast measured by 7-point Likert Scales | 2 times: 0-12h fasting- and 15 minutes after breakfast consumption
  healthy, satiating, palatable, energizing and caloric perception
Self-reported appetite and satiety ratings measured by Visual Analog rating Scales | 0-12h fasting- and every 30 minutes up to 4 hours after breakfast consumption
Food choices at subsequent meal measured by double weighing of food during an ad libitum lunch buffet | 4 hours after breakfast conusmption
Daily Energy Intake measured by 7-day food dairy | 7 days
  Energy intake during breakfast, morning snacks, lunch, afternoon snacks, dinner, and evening snacks
Post-prandial attention measured by Mackworth Clock Test and Stroop Test | 4 hours after breakfast conusmption
  sustained and selective attention
Brain activation responses to images of food measured by fMRI brain scan | 4 hours after breakfast conusmption

CONTACTS AND LOCATIONS:
Overall Officials: Furio Brighenti, Professor, Principal Investigator — University of Parma
Locations (1):
- University of Parma, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rosi A, Martini D, Scazzina F, Dall'Aglio E, Leonardi R, Monti L, Fasano F, Di Dio C, Riggio L, Brighenti F. Nature and Cognitive Perception of 4 Different Breakfast Meals Influence Satiety-Related Sensations and Postprandial Metabolic Responses but Have Little Effect on Food Choices and Intake Later in the Day in a Randomized Crossover Trial in Healthy Men. J Nutr. 2018 Oct 1;148(10):1536-1546. doi: 10.1093/jn/nxy160. PMID 30204905